CLINICAL TRIAL: NCT03340298
Title: The Effect of a Weight Reducing Diet Containing Different Sources of Fiber on Cardiovascular Risk Factors in Overweight and Obese Women: A Randomized Feeding Trial
Brief Title: Fiber and Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIBER
Record Dates: First submitted 2017-11-05; First posted 2017-11-13 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- grain (Experimental): 25 gram fiber from whole grain products and 10 gram fiber from fruits and vegetables
  Interventions: Dietary Supplement: fiber
- fruits and vegetables (Experimental): 25 gram fiber from fruits and vegetables as main supplier and the remaining 10 grams from whole grain sources
  Interventions: Dietary Supplement: fiber
- grain-fruits and vegetables (Experimental): 17.5 gram fiber from whole grain and 17.5 gram fiber from fruits and vegetables
  Interventions: Dietary Supplement: fiber

INTERVENTIONS:
Dietary Supplement: fiber — the intervention of different sources of dietary fibers

SUMMARY:
This study was a parallel randomized controlled feeding trial conducted in overweight and obese participants who were attending the Nutrition Clinic in Isfahan, Iran. Inclusion criteria were as follows: women aged 18 to 50 years; body mass index (BMI) 25 kg/m2

; having noncommunicable diseases such as diabetes, hyperlipidemia, and hypertension; having no history of liver and renal disease, hormonal disorders, food allergy, and other special diseases; not taking specific medications affecting weight; willingness to introduce a dietary change to lose weight; and habitual daily consumption of fruits, vegetables, and whole grains. The exclusion criteria were the following: weight loss of more than 10% of body weight within the 6 months before registration in the study; attending a competitive sport; no consumption of fruits, vegetables, or whole grains habitually; abnormal thyroid hormone concentration; intake of drugs or supplementation that could affect energy expenditure or weight; and not following recommended diets or returning for following visits. Recruitment ran from January 2016 to July 2016. The sample size was calculated based on the standard formula (45):

by considering the Type 1 error (a) of 0.05 and Type 2 error (b) of 0.20 (power D 80%). Based on a previous study in Iranian women (46), we used a within-group BMI mean difference (d) of 2.5 kg/m2 and a standard deviation (SD) of 3.2 kg/m2

* Therefore, we needed 25 participants in each group. The study was approved by the research council and ethical committee of the School of Nutrition and Food Science, Isfahan University of Medical Sciences, Isfahan, Iran (grant number: 194172). All participants gave written consent before study enrollment. This trial was registered at ClinicalTrial.gov with code NCT03340298. Study design and interventions A randomized feeding trial was designed that aimed to compare the effect of different sources of fibers with low-calorie conventional diets on weight loss, waist circumference (WC), blood pressure, fasting blood glucose (FBS), and lipid profiles in overweight and obese women. Eligible participants were randomly assigned to the three groups after baseline measures of BMI, using a computer-generated random numbers method of randomization. Seventy-five participants who were eligible for the study were randomly divided to one of the three groups ("whole grains" high fiber diet, "fruits and vegetables" high fiber diet, and diet containing "whole grains, fruits, and vegetables") in a 1:1:1 allocation (Figure 2). Participant allocation was stratified by age and BMI. All participants consumed 35 g of fiber per day as follows: in the whole grains group (n D 25), 25 g of fiber from whole grain products and 10 g fiber from fruits and vegetables was to be consumed with the main meals; in the fruits and vegetables group (n D 25), 25 g of fiber from fruits and vegetables and 10 g from whole grain sources was to be consumed with the main meals; and in the whole grains, fruits, and vegetables group, participants were to consume an equal amount of fiber from both sources (17.5 g fiber from whole grains and 17.5 g fiber from fruits and vegetables) with their main meals daily for 10 weeks. The main meals were determined by an expert dietitian, based on the Harris-Benedict formula, considering 0.5 kg weekly weight loss for each participant. The distribution of macronutrients was similar among groups (carbohydrates, 55%; fat, 30%; and protein, 15%) and the number of servings of each food group was estimated and given to participants. Participants in each group were given their allowed food that contained a list of exchangeable foods, food groups, and subgroups (Table 2). All participants were instructed to attend the nutrition clinic to take their intended products. Participants were supplied with the fruits, vegetables, and whole grains for their diet and they consumed these food items under supervision in the nutrition clinic for 10 weeks. Other components of their weight loss diets, such as dairy, meats/alternatives, and fat groups were asked to be consumed in a free-living situation. To assess compliance of participants' intake of weight loss diets, participants were asked to record their 24-hour food intakes for 3 d/wk during weeks 2, 5, and 10 of the trial. Duration of all physical activities was collected, similar to dietary intakes. To obtain the metabolic equivalent for daily physical activity, the recorded physical activities were multiplied by the relevant metabolic equivalents task hours per day (MET-h/d) to give the MET-h/d values.

ELIGIBILITY:
Inclusion Criteria:

overweight or obese

Exclusion Criteria:

have any diseases

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — the overweight or obese female that referred to the Clinic Nutrition to lose weight
Enrollment: 75 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
change of weight | 10 weeks
  Weight was measured by using a digital scale to the nearest 100g while participants wearing light clothes ( Seca, Hamburg , Germany)

SECONDARY OUTCOMES:
change of waist circumference | 10 weeks
  The narrowest part of Waist was considered for measuring waist circumference where is between the last rib and the iliac crest to the nearest 0.1 cm over light clothing .

OTHER OUTCOMES:
change of BMI | 10 weeks
  BMI was calculated as body weight (Kg)/ height 2 (m).We used a standard mercury sphygmomanometer to measure participants
change of blood pressure | 10 weeks
  Blood pressure after resting for 15 minutes. The measurement was performed three times in the sitting position with 1 minute intervals and the average of three measurements was considered as final blood pressure.Systolic blood pressure was defined as the appearance of the first sound and diastolic blood pressure was defined as the disappearance of the sound.(Korotkoff phase 5).All Subjects were asked to avoid coffee, tea and all caffeine containing materials before blood pressure.
change of FBS | 10 weeks
  Fasting blood glucose was measured by enzymatic colorimetric method using glucose oxidase on the day of blood collection.Blood Specimens were centrifuged at 3000 rpm for 10 minutes in order to separate plasma and samples were stored at -70 C until analysis
change of lipid profiles | 10 weeks
  Total cholesterol level and serum TG analysis was done using a Selectra 2 auto-analyzer (Vital scientific, Spankeren ,The Netherlands.) by an enzymetic colorimetric method with cholesterol esterase and cholesterol oxidase and glycerol phosphate oxidase.(Parsazmoun,Tehran ,Iran). HDL-C determination was done after precipitation of apolipoprotein B containing lipoporotein withphosphotungstic acid. LDL-C was calculated by Friedewald ´s formula when the TAG level was lower than 400 mg/dl ; otherwise , LDL-C was determined by an enzymatic method